CLINICAL TRIAL: NCT06431451
Title: The Correlation Between Ripretinib Exposure and the Efficacy and Safety in Patients with Advanced Gastrointestinal Stromal Tumors: an Observational Study
Brief Title: The Correlation Between Ripretinib Exposure and the Efficacy and Safety in Patients with Advanced GISTs
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xinhua Zhang, MD, Chief physician, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 20240102v3.0
Record Dates: First submitted 2023-12-24; First posted 2024-05-28 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-05

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Ripretinib; plasma drug concentration
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, single-center, observational study to explore the correlation between ripretinib exposure and the efficacy and safety in patients with advanced gastrointestinal stromal tumors

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE:

Gastrointestinal stromal tumors (GISTs) are a rare mesenchymal sarcoma that most commonly occur in the stomach and small intestine, but can occur in any region of the entire gastrointestinal tract. For advanced GISTs that cannot be surgically removed or metastasized, imatinib, sunitinib, and regorafenib are recommended TKIs in the current clinical guidelines for the first-, second-, and third-line therapy respectively. Although imatinib has significant effect in the first-line treatment of GIST, improving the prognosis and survival outcome, GISTs often develop primary or secondary drug resistance, resulting in disease progression.Ripretinib is a broad-spectrum switch-control kinase inhibitor that specifically inhibits KIT and PDGFRA kinase signaling through dual mechanisms of action. In clinical studies of advanced GIST patients, Ripretinib has shown good safety and efficacy. In the phase III clinical study INVICTUS, Ripretinib 150 mg QD was used to treat patients with metastatic or unresectable GIST who failed to treatment with imatinib, sunitinib, and regorafenib. The median progression-free survival (mPFS) was 6.3 months in the Ripretinib group and 1.0 month in the placebo group. The phase III clinical trial INTRIGUE showed that although there was no significant advantage in progression-free survival (PFS) compared with sunitinib, Ripretinib had better safety, lower incidence of adverse events, and better patient tolerability. In May 2020, Ripretinib was approved by the US FDA for the treatment of adult patients with advanced GIST who have failed to three or more kinase inhibitors including imatinib. It is also recommended as a preferred fourth-line drug in the 2023 version of the NCCN guidelines and the 2022 version of the CSCO guidelines for GISTs.

In vitro kinase and cell studies have shown that Ripretinib is effective against wild-type KIT and PDGFRA, as well as a wide range of KIT and PDGFRA mutations, including major and resistant mutations in KIT exons 9, 11, 13, 14, 17, and 18, as well as the regorafenib-resistant D816V mutation. It is more effective than other type I and type II TKI inhibitors. However, the inhibitory effect of Ripretinib varies depending on the mutation type. At the same time, in the phase III clinical study INVICTUS gene mutation analysis, it was found that patients with primary mutations in KIT exon 11 and secondary mutations in KIT exon 17 had a relatively longer PFS.

The preclinical study of Ripretinib suggests that its inhibitory effect on KIT is concentration-dependent and time-dependent. With the increase of in vivo concentration, the inhibitory effect of KIT phosphorylation also increases. Increasing the dosage or dosing frequency can increase tumor regression and survival rates. In the phase I clinical study of Ripretinib, it was found that increasing the dose to 150 mg BID after oral administration of 150mg QD with disease progression (PD) can obtain a further benefit. The median progression-free survival (mPFS) of second-line, third-line, and fourth-line patients was 5.6, 3.3, and 4.6 months, respectively, indicating that the increase of Ripretinib's exposure in vivo is associated with improved efficacy.

Preclinical and clinical studies have found that the main metabolic pathway of Ripretinib is N-demethylation. Ripretinib and its active metabolite DP-5439 are mainly metabolized in the liver through CYP3A4 metabolic enzymes, and DP-5439 has pharmacological activity similar to the parent drug Ripretinib. In a phase I clinical study of pharmacokinetics, there was significant inter-patient variability in PK parameters after administration of Ripretinib. The variation (CV%) of Cmax and AUC0-24h reached 35% to 60%. The AUC of DP-5439 after a single dose of 150 mg was about 49% of Ripretinib, and the AUC after 15 days of dosing at 150 mg QD was about 129% of Ripretinib. At the same time, the AUC0-24h of Ripretinib increased proportionally with dose within the range of 20-250 mg, but the Cmax increased less than dose proportionally. The Cmax and AUC0-24h of DP-5439 increased less than dose proportionally within the range of 50-250 mg.The above findings suggest that therapeutic drug monitoring (TDM) may be clinically relevant for patients receiving Ripretinib treatment, and further exploration of the relationship between blood concentration or exposure level of Ripretinib and clinical efficacy is warranted.

In terms of safety, in the phase I dose-escalation trial of Ripretinib, no maximum tolerated dose (MTD) was found, and the dose-limiting toxicity (DLT) was elevation of lipase and creatine kinase, which occurred in dose groups of 100 mg BID, 200 mg BID, and 150 mg QD. The most common treatment-related adverse events included fatigue, alopecia, nausea, muscle pain, constipation, loss of appetite, palmoplantar erythrodysesthesia syndrome (PPES), diarrhea, and elevation of lipase. Most of these events were mild to moderate. The incidence of serious adverse events was 14.1%, including elevation of creatine kinase, elevation of lipase, elevation of bilirubin, myocardial infarction, and heart failure. In the phase I dose-escalation trial, it was shown that the incidence of adverse events such as muscle pain, muscle spasms, PPES, and hypertension increased with dose escalation, indicating a possible dose-related toxicity. Therefore, in order to reduce the occurrence of adverse reactions and improve medication safety, it is of great significance to find a relatively safe dose range to guide clinical safe drug use.

In addition, although the results of the phase II clinical trial of Ripretinib in China suggested that the efficacy, safety, and PK characteristics of Ripretinib in Chinese patients were consistent with the global patient population, a comparison of the results between Chinese patients and global patients in the phase I clinical trial showed that the clinical efficacy of Chinese patients receiving Ripretinib as a fourth-line treatment at a dose of 150 mg QD was slightly better than that of global patients (mPFS: 7.2 vs. 6.3 months; ORR: 18.4% vs. 11.8%). Meanwhile, the overall exposure of Ripretinib and DP-5439 was slightly higher in the Chinese population compared to global data. This suggests that it is worth further exploring the relationship between the pharmacokinetics and exposure of Ripretinib in the Chinese population and its efficacy, which has implications for personalized treatment in Chinese patients.

This study aims to establish a method for monitoring the blood concentrations of Ripretinib and its active metabolite DP-5439, and to monitor the blood concentrations of advanced GIST patients receiving Ripretinib treatment. The study will explore the relationship between the exposure of Ripretinib and its efficacy and safety in real-world advanced GIST patients, determine the therapeutic window of Ripretinib, and explore the effective exposure levels required for different KIT mutation types.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged ≥ 18 years.
* Gastrointestinal stromal tumors confirmed by histopathological examination, and CD117 and/or DOG-1-positive by immunohistochemistry.
* patients who are currently receiving Ripretinib treatment.
* Subjects must have at least one measurable lesion based on mRECIST v1.1 criteria, and have undergone at least one radiographic evaluation for efficacy analysis.
* Patients with an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 4
* Patient informed consent and signed written consent form.
* The patient was compliant and voluntarily scheduled for follow-up, treatment, laboratory tests, and other study procedures.

Exclusion Criteria:

* Unable to complete at least 15 consecutive days of Ripretinib due to intolerance or disease progression.
* Individuals with other serious acute or chronic physical or mental health problems, or abnormal laboratory test results that increase the risk associated with participation in the study or use of the drug, or that could interfere with the interpretation of study results, and who, in the opinion of the investigator, are not suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastrointestinal stromal tumor patients who are receiving treatment with Ripretinib at the research center.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of ripretinib | Before Dosing and at 0.5, 1, 2, 4, 6, 8,12 and 24 Hours after Dosing
  The concentration of ripretinib in the plasma was measured.
Plasma Concentration of DP-5439 | Before Dosing and at 0.5, 1, 2, 4, 6, 8,12 and 24 Hours after Dosing
  The concentration of DP-5439 in the plasma was measured.
Objective Response Rate | 2 years
  To evaluate objective response rate (ORR,CR+PR) determined by radiology assessment per mRECIST(Response Evaluation Criteriain Solid Tumours), version 1.1 in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.Complete response is the disappearance of all lesions with lymph nodes measuring < 10 mm and normal tumour markers.A decrease in the sum of target disease of ≥ 30% represents partial response.
Disease control rate | 2 years
  To evaluate disease control rate (CBR,CR+PR+>16 weeks continuation SD) determined by radiology assessment per mRECIST, version 1.1 in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.Complete response is the disappearance of all lesions with lymph nodes measuring < 10 mm and normal tumour markers.A decrease in the sum of target disease of ≥ 30% represents partial response.Stable disease lies between partial response and progressive disease.

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  Progression-free survival (PFS) is defined as the interval between the date of drug administration and the earliest date of disease progression or death due to any cause.
overall survival | 2 years
  Overall survival is defined as the time from drug administration until death.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] von Mehren M, Joensuu H. Gastrointestinal Stromal Tumors. J Clin Oncol. 2018 Jan 10;36(2):136-143. doi: 10.1200/JCO.2017.74.9705. Epub 2017 Dec 8. PMID 29220298
- [Background] Di Vito A, Ravegnini G, Gorini F, Aasen T, Serrano C, Benuzzi E, Coschina E, Monesmith S, Morroni F, Angelini S, Hrelia P. The multifaceted landscape behind imatinib resistance in gastrointestinal stromal tumors (GISTs): A lesson from ripretinib. Pharmacol Ther. 2023 Aug;248:108475. doi: 10.1016/j.pharmthera.2023.108475. Epub 2023 Jun 10. PMID 37302758
- [Background] Zalcberg JR. Ripretinib for the treatment of advanced gastrointestinal stromal tumor. Therap Adv Gastroenterol. 2021 Apr 15;14:17562848211008177. doi: 10.1177/17562848211008177. eCollection 2021. PMID 33948116
- [Background] Janku F, Abdul Razak AR, Chi P, Heinrich MC, von Mehren M, Jones RL, Ganjoo K, Trent J, Gelderblom H, Somaiah N, Hu S, Rosen O, Su Y, Ruiz-Soto R, Gordon M, George S. Switch Control Inhibition of KIT and PDGFRA in Patients With Advanced Gastrointestinal Stromal Tumor: A Phase I Study of Ripretinib. J Clin Oncol. 2020 Oct 1;38(28):3294-3303. doi: 10.1200/JCO.20.00522. Epub 2020 Aug 17. PMID 32804590
- [Background] Smith BD, Kaufman MD, Lu WP, Gupta A, Leary CB, Wise SC, Rutkoski TJ, Ahn YM, Al-Ani G, Bulfer SL, Caldwell TM, Chun L, Ensinger CL, Hood MM, McKinley A, Patt WC, Ruiz-Soto R, Su Y, Telikepalli H, Town A, Turner BA, Vogeti L, Vogeti S, Yates K, Janku F, Abdul Razak AR, Rosen O, Heinrich MC, Flynn DL. Ripretinib (DCC-2618) Is a Switch Control Kinase Inhibitor of a Broad Spectrum of Oncogenic and Drug-Resistant KIT and PDGFRA Variants. Cancer Cell. 2019 May 13;35(5):738-751.e9. doi: 10.1016/j.ccell.2019.04.006. PMID 31085175
- [Background] Klug LR, Khosroyani HM, Kent JD, Heinrich MC. New treatment strategies for advanced-stage gastrointestinal stromal tumours. Nat Rev Clin Oncol. 2022 May;19(5):328-341. doi: 10.1038/s41571-022-00606-4. Epub 2022 Feb 25. PMID 35217782
- [Background] Blay JY, Serrano C, Heinrich MC, Zalcberg J, Bauer S, Gelderblom H, Schoffski P, Jones RL, Attia S, D'Amato G, Chi P, Reichardt P, Meade J, Shi K, Ruiz-Soto R, George S, von Mehren M. Ripretinib in patients with advanced gastrointestinal stromal tumours (INVICTUS): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2020 Jul;21(7):923-934. doi: 10.1016/S1470-2045(20)30168-6. Epub 2020 Jun 5. PMID 32511981
- [Background] Bauer S, Jones RL, Blay JY, Gelderblom H, George S, Schoffski P, von Mehren M, Zalcberg JR, Kang YK, Razak AA, Trent J, Attia S, Le Cesne A, Su Y, Meade J, Wang T, Sherman ML, Ruiz-Soto R, Heinrich MC. Ripretinib Versus Sunitinib in Patients With Advanced Gastrointestinal Stromal Tumor After Treatment With Imatinib (INTRIGUE): A Randomized, Open-Label, Phase III Trial. J Clin Oncol. 2022 Dec 1;40(34):3918-3928. doi: 10.1200/JCO.22.00294. Epub 2022 Aug 10. PMID 35947817
- [Background] Li J, Cai S, Zhou Y, Zhang J, Zhou Y, Cao H, Wu X, Deng Y, Huang Z, Dong J, Shen L. Efficacy and Safety of Ripretinib in Chinese Patients with Advanced Gastrointestinal Stromal Tumors as a Fourth- or Later-Line Therapy: A Multicenter, Single-Arm, Open-Label Phase II Study. Clin Cancer Res. 2022 Aug 15;28(16):3425-3432. doi: 10.1158/1078-0432.CCR-22-0196. PMID 35686969
- [Background] George S, Chi P, Heinrich MC, von Mehren M, Jones RL, Ganjoo K, Trent J, Gelderblom H, Razak AA, Gordon MS, Somaiah N, Jennings J, Meade J, Shi K, Su Y, Ruiz-Soto R, Janku F. Ripretinib intrapatient dose escalation after disease progression provides clinically meaningful outcomes in advanced gastrointestinal stromal tumour. Eur J Cancer. 2021 Sep;155:236-244. doi: 10.1016/j.ejca.2021.07.010. Epub 2021 Aug 12. PMID 34391056
- [Background] Zalcberg JR, Heinrich MC, George S, Bauer S, Schoffski P, Serrano C, Gelderblom H, Jones RL, Attia S, D'Amato G, Chi P, Reichardt P, Somaiah N, Meade J, Reichert V, Shi K, Sherman ML, Ruiz-Soto R, von Mehren M, Blay JY. Clinical Benefit of Ripretinib Dose Escalation After Disease Progression in Advanced Gastrointestinal Stromal Tumor: An Analysis of the INVICTUS Study. Oncologist. 2021 Nov;26(11):e2053-e2060. doi: 10.1002/onco.13917. Epub 2021 Aug 16. PMID 34313371
- [Background] Pan C, Cheng Y, He Q, Li M, Bu F, Zhu X, Li X, Xiang X. Evaluating the impact of co-administered drug and disease on ripretinib exposure: A physiologically-based pharmacokinetic modeling approach. Chem Biol Interact. 2023 Mar 1;373:110400. doi: 10.1016/j.cbi.2023.110400. Epub 2023 Feb 9. PMID 36773833
- [Background] Li X, Shelton MJ, Wang J, Meade J, Ruiz-Soto R. Effects of CYP3A Inhibition, CYP3A Induction, and Gastric Acid Reduction on the Pharmacokinetics of Ripretinib, a Switch Control KIT Tyrosine Kinase Inhibitor. Clin Pharmacol Drug Dev. 2022 Oct;11(10):1165-1176. doi: 10.1002/cpdd.1110. Epub 2022 May 13. PMID 35560823
- [Background] Demetri GD, Wang Y, Wehrle E, Racine A, Nikolova Z, Blanke CD, Joensuu H, von Mehren M. Imatinib plasma levels are correlated with clinical benefit in patients with unresectable/metastatic gastrointestinal stromal tumors. J Clin Oncol. 2009 Jul 1;27(19):3141-7. doi: 10.1200/JCO.2008.20.4818. Epub 2009 May 18. PMID 19451435
- [Background] Yang W, Qian H, Yang L, Wang P, Qian H, Chu B, Liu Z, Sun J, Wu D, Sun L, Zhou W, Hu J, Chen X, Shou C, Ruan L, Zhang Y, Yu J. Efficacy and safety of ripretinib in Chinese patients with advanced gastrointestinal stromal tumors: a real-world, multicenter, observational study. Front Oncol. 2023 May 18;13:1180795. doi: 10.3389/fonc.2023.1180795. eCollection 2023. PMID 37274264